CLINICAL TRIAL: NCT01190280
Title: Indications for Gallbladder Surgery in Gallstone Disease
Status: Completed | Type: Observational
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Karl Søndenaa, Haraldsplass Deaconal Hospital, Department of Surgery, University of Bergen, Bergen, Norway
Other Study IDs: GS06
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-08

CONDITIONS: Gallstones
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — Resected gallbladders for histological and bacteriological investigation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- AC - operation: Patients admitted with acute cholecystitis randomized to operation
  Interventions: Procedure: Cholecystectomy operation
- AC - observation: Patients admitted with acute cholecystitis randomized to observation
- SGBS - operation: Patients admitted with uncomplicated gallstone disease randomized to operation
  Interventions: Procedure: Cholecystectomy operation
- SGBS - observation: Patients admitted with uncomplicated gallstone disease randomized to observation
- 1983 - stones: Patients that in 1983 were diagnosed with gallstones in a population screening
- 1983 - operation: Patients that were operated for gallstone disease at Haukeland University Hospital, Bergen, Norway, in 1983
- 1983 - controls: Patients that were shown not to have gallstones in a 1983 population screening
- Gallstone patients: Patients with symptoms from gallstone disease

INTERVENTIONS:
Procedure: Cholecystectomy operation — Cholecystectomy after randomization
  Other Names: Removal of gallbladder
  Groups: AC - operation; SGBS - operation

SUMMARY:
The aim of the study is to identify patients with gallstone disease that should be operated and those that may potentially be observed. This selection was based on symptoms and clinical presentation. The consequences that may arise for the patient if observation is chosen compared with outcome after cholecystectomy has been markers of outcome.

DETAILED DESCRIPTION:
1. Randomized clinical trial (RCT) of observation versus surgery for uncomplicated gallstone disease
2. RCT of observation versus operation for acute cholecystitis
3. Study of outcome after cholecystectomy in patients from 1. and 2.
4. Study of symptoms in gallstone disease and symptom relief after cholecystectomy
5. Long-term morbidity and mortality, including cancer, after cholecystectomy
6. Long-term follow-up of patients with silent gallstones

ELIGIBILITY:
Inclusion criteria:

* Symptomatic gallstone disease (SGBS):

Episodes of pain in the right subcostal or midline epigastric area lasting more than 30 min, with ultrasonography signs of gallstones.

* Ultrasonographic: echo with an acoustic shadow in a visible gallbladder, or an echo with positional change and size <3 mm or, alternatively no demonstrable gallbladder but a strong echo with an acoustic shadow in the position of the gallbladder

Exclusion Criteria SGBS:

* Infrequent and/or minimal pain that need only very occasional medication
* Age below 18 or above 80
* Not willing to participate

Inclusion criteria, acute cholecystitis (AC):

* Acute abdominal pain
* Duration of more than 8-12 h
* Tenderness on clinical examination in the upper right quadrant
* Presence of gallbladder stones and signs of inflammation on ultrasonography and in clinical biochemistry data, including an elevated temperature

Exclusion criteria, AC:

* Severe concomitant disease
* Suspected Common Bile Duct stone
* Acalculous cholecystitis
* Localized peritonitis suggesting gallbladder perforation or gangrenous cholecystitis

Inclusion criteria 1983 cohort of patients:

* Participation in a screening study for gallstones in 1983
* Operated for symptomatic gallstone disease in Bergen, Norway in 1983

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a hospital for either acute cholecystitis or uncomplicated symptomatic gallstone disease randomized to observation or operation. Patients from a population screening study for gallstones performed in 1983. Patients operated for gallstone disease in 1983.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 1991-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl Søndenaa, MD, PhD, Study Chair — Haraldsplass Deaconal Hospital, University of Bergen, Norway
Locations (1):
- Haraldsplass Deaconal Hospital, Department of Surgery, Bergen, Norway

REFERENCES:
- [Background] Sondenaa K, Nesvik I, Solhaug JH, Soreide O. Randomization to surgery or observation in patients with symptomatic gallbladder stone disease. The problem of evidence-based medicine in clinical practice. Scand J Gastroenterol. 1997 Jun;32(6):611-6. doi: 10.3109/00365529709025108. PMID 9200296
- [Background] Glambek I, Kvaale G, Arnesjo B, Soreide O. Prevalence of gallstones in a Norwegian population. Scand J Gastroenterol. 1987 Nov;22(9):1089-94. doi: 10.3109/00365528708991963. PMID 3321395
- [Background] Vetrhus M, Soreide O, Solhaug JH, Nesvik I, Sondenaa K. Symptomatic, non-complicated gallbladder stone disease. Operation or observation? A randomized clinical study. Scand J Gastroenterol. 2002 Jul;37(7):834-9. PMID 12190099
- [Background] Vetrhus M, Soreide O, Nesvik I, Sondenaa K. Acute cholecystitis: delayed surgery or observation. A randomized clinical trial. Scand J Gastroenterol. 2003 Sep;38(9):985-90. doi: 10.1080/00365520310004056. PMID 14531537
- [Background] Vetrhus M, Berhane T, Soreide O, Sondenaa K. Pain persists in many patients five years after removal of the gallbladder: observations from two randomized controlled trials of symptomatic, noncomplicated gallstone disease and acute cholecystitis. J Gastrointest Surg. 2005 Jul-Aug;9(6):826-31. doi: 10.1016/j.gassur.2005.01.291. PMID 15985239
- [Derived] Schmidt M, Smastuen MC, Sondenaa K. Increased cancer incidence in some gallstone diseases, and equivocal effect of cholecystectomy: a long-term analysis of cancer and mortality. Scand J Gastroenterol. 2012 Dec;47(12):1467-74. doi: 10.3109/00365521.2012.719928. Epub 2012 Sep 5. PMID 22946484